CLINICAL TRIAL: NCT04326075
Title: EC-COVID-RCT. Early CPAP in COVID Patients With Respiratory Failure. A Randomized Clinical Trial
Brief Title: Early CPAP in COVID-19 Patients With Respiratory Failure.
Acronym: EC-COVID-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-COVID-RCT-Fenice
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2021-12

CONDITIONS: CPAP Ventilation; COVID-19; Emergency Departments
MeSH Terms: conditions — COVID-19; Emergencies | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early CPAP treatment (Experimental): Early treatment with CPAP in addition to current clinical practice
  Interventions: Device: CPAP treatment
- Control (No Intervention): Current clinical practice, which currently does not involve the use of CPAP.

INTERVENTIONS:
Device: CPAP treatment — CPAP should be performed as soon as possible and only with a helmet, using a positive end-expiratory pressure (PEEP) between 8 and 14 cmH2O and an inspired oxygen fraction (FiO2) between 40 and 60%.
  Arms: Early CPAP treatment

SUMMARY:
The study aims at clarifying whether early treatment with continuous positive airway pressure (CPAP) ventilation is able to reduce the need for intubation or death in patients visiting an emergency department (ED) with known or suspected COVID-19 infection and insufficiency respiratory.

DETAILED DESCRIPTION:
Eligible patients will be randomized to two treatment arms: current clinical practice (control arm) and early treatment with CPAP in addition to current clinical practice (experimental arm). To deal with the current emergency situation, the study will adopt an adaptive design with a Bayesian continuous monitoring. Such design allows to stop the study as soon as the data provide sufficient evidence of efficacy or ineffectiveness of the studied treatment.

The primary endpoint of the study is the combination of intubation or death within 7 days of randomization. The secondary endpoint is 30-day mortality.

All patients arriving at the ED will be evaluated to verify the presence of inclusion and exclusion criteria. Randomization will be performed through an ad-hoc electronic case report form (eCRF). Eligible patients should be randomized as soon as possible, possibly immediately after the ED triage.

Patients randomized to the control arm will be treated according to current clinical practice, which currently does not involve the use of CPAP. Therefore, these patients should not start treatment with CPAP immediately after randomization. CPAP treatment, however, is allowed at a later stage, if deemed appropriate according to clinical judgment.

Patients randomized to the experimental arm should begin treatment with CPAP as soon as possible. CPAP should only be performed with a helmet, using a positive end-expiratory pressure (PEEP) between 8 and 14 cmH2O and an inspired oxygen fraction (FiO2) between 40 and 60%. FiO2 and PEEP must be modulated, within the limits indicated above, so as to obtain a saturation > 94%. Whenever this goal cannot be achieved, the patient should be referred to the intensivist.

ELIGIBILITY:
Inclusion Criteria:

ED patients positive to or suspected of COVID-19 infection with at least one of the following symptoms:

* fever
* cough/dyspnea
* respiratory symptoms or ED arrival for respiratory reason and for whom there are the following conditions:
* SpO2 < 95% in ambient air or positive Quick Walk Test
* PaO2/FiO2 > 200 in ambient air or with Venturi mask, evaluated in 1 hour from ED arrival.

Exclusion Criteria:

* BPCO patients
* Age > 70 years
* Pregnant status
* Contraindications for CPAP

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Death or need of intubation | 7 days since ED arrival
  The study outcomes will be death or need of intubation within 7 days since ED arrival.

SECONDARY OUTCOMES:
30-day mortality | 30 days since ED arrival
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided